CLINICAL TRIAL: NCT04677920
Title: The HEALTHY COOKIE ENERGY STUDY: Understanding How Healthy Cookies Affect Mitochondrial Biology
Acronym: HCES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0352
Record Dates: First submitted 2020-09-18; First posted 2020-12-21 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Cookie Group (Experimental): All participants in the study
  Interventions: Other: High Linoleic Acid Healthy Cookies

INTERVENTIONS:
Other: High Linoleic Acid Healthy Cookies — High Linoleic Acid Healthy Cookies (containing about 10g of grapeseed oil) 1 per day for 2 weeks

SUMMARY:
The proposed research is an intervention and feasibility pilot trial designed to determine if short-term consumption of healthy cookies made with an oil rich in linoleic acid can influence mitochondria biology in white blood cells and muscle. The hypothesis of the study is that consuming 1 healthy cookie rich in linoleic acid each day for two weeks will improve mitochondrial biology in white blood cells and muscle.

DETAILED DESCRIPTION:
Linoleic acid has many health benefits including altering body composition and energy metabolism, possibly through its impact on cardiolipin and mitochondria.

The investigators plan to test the central hypothesis and accomplish the overall objective of this research by pursuing the following four specific aims

Aim 1) To assess muscle biopsy yield with a micro biopsy needle

Aim 2) To determine the amount of peripheral blood mononuclear cells (PBMC) and muscle needed to measure mitochondria function

Aim 3) To assess the feasibility of measuring mitochondria function on fresh PBMC and muscle samples

Aim 4) To determine the effect of short-term healthy cookies made with linoleic acid rich oil on measures of mitochondrial function in white blood cells and muscle as well as their relationship to lipid composition of the blood, markers of metabolic health and markers of mitochondria biogenesis

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker

Exclusion Criteria:

* Allergy/intolerance to lidocaine
* Gastrointestinal diseases or disorders (including pancreatic) or gastric bypass surgery
* Food Allergy or Intolerance
* Any dietary restriction where consumption of these healthy cookies or any ingredient would be contraindicated
* Use of medications where consuming the healthy cookies would be contraindicated
* Pregnancy
* Use of anticoagulant, antiplatelet, or other blood thinner medications
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in mitochondria function | Week 0 to Week 2
  Mitochondria function measured in peripheral blood mononuclear cells and skeletal muscle
Changes in cardiolipin species | Week 0 to week 2
  Cardiolipin species in peripheral blood mononuclear cells and skeletal muscle
Correlation of mitochondrial biology in blood and skeletal muscle | Week 0 and week 2
  Correlation of mitochondria function and cardiolipin species in peripheral blood mononuclear cells and skeletal muscle

SECONDARY OUTCOMES:
Changes in fasting fatty acid levels | Week 0 to week 2
  Linoleic acid content of fasting blood samples
Correlation of fatty acids with mitochondrial function and cardiolipin species | Week 0 and week 2
  Correlation of linoleic acid in blood with mitochondria function and cardiolipin species in peripheral blood mononuclear cells and skeletal muscle
Correlation of cardiolipin with global sleep quality score, Cambridge physical activity index and dietary intake of omega-3 fats | Week 0 and week 2
  Correlation of cardiolipin in peripheral blood mononuclear cells and skeletal muscle with measurements of sleep quality using the Pittsburgh Sleep Quality Index, physical activity using the Epic Physical activity short questionnaire and dietary omega-3 intake using the Omega-3 Checklist
Correlation of cardiolipin with body mass index, sagittal diameter (abdominal thickness), walking speed and grip strength | Week 0 and week 2
  Correlation of cardiolipin in peripheral blood mononuclear cells and skeletal muscle with measurements of body mass index, sagittal diameter, grip strength and gait speed

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No